CLINICAL TRIAL: NCT05434715
Title: Evaluation of Minimal Invasive Thyroidectomy; A Randomized Controlled Trial
Brief Title: Evaluation of Minimal Invasive Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Aouf, Dr, assistant lecturer of General Surgery, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MKSU50-6-19
Record Dates: First submitted 2022-06-20; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Thyroid; Goiter
MeSH Terms: conditions — Thyroid Diseases; Goiter | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional technique of thyroidectomy (Active Comparator): A standard transverse skin incision will be done two fingers above supra-sternal notch extend from the medial head of sternomastoid muscle at one side to the other one at the opposite side, incision of platysma along the whole length of skin incision.
  Dissection of the thyroid gland will begin with securing the middle thyroid vein using ligation, bipolar diathermy, or harmonic scalpel.
  Dissection of the upper pole with securing the superior thyroid vessel preserving the superior parathyroid glands and the external laryngeal nerve.
  Severing the Berry's ligament with ligation of its artery and vein. The contralateral lobe of the thyroid gland will then be approached in a similar fashioon.
  Interventions: Procedure: Thyroidectomy
- Minimal invasive technique (Active Comparator): The procedure will start by placing a small incision 2.5-3cm at the upper border of the cricoid cartilage at one of the natural creases of the neck, followed by an incision of the platysma along the length of the skin incision.
  Identification of the midline of the neck and division of the strap muscles, followed by dissection of the plane between the muscles and the anterior surface of the thyroid gland.
  Dissection of the lateral surface of the thyroid lobe with identification Cutting of sternothyroid muscle at its superior portion. Individual ligaton of branches of superior thyroid artery and vein near to the gland using haemostatic techniques (Harmonic or LigaSure scalpel), guarding the superior parathyroid glands.
  Appropriate dissection will then be done. Dissection of the inferior pole and vessel securing using Harmonic or LigaSure scalpel will take place, then dissection of the undersurface of the thyroid gland will be done to separate the gland from its bed.
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — removal of the thyroid gland

SUMMARY:
The goals of minimally invasive approaches are better cosmetic results with small neck scar, decreasing postoperative pain, and shortening of hospital stay periods without postoperative complications.

The concept of surgical invasiveness cannot be limited to the length and site of the skin incision; it must be extended to all structures dissected during the procedure. Conventional thyroidectomy without raising subplatysmal flaps has proven to be effective in reducing postoperative pain and seroma

DETAILED DESCRIPTION:
Minimal invasive flapless thyroidectomy (MIFT) is a new technique that can be used in replacement of the conventional method of thyroidectomy for the management of selected cases of benign thyroid disorders.

This work aims to evaluate the feasibility, safety, and efficacy of Minimal Invasive Flapless Thyroidectomy (MIFT) in the management of thyroid disease as regards postoperative pain, cosmesis, operative time, and other postoperative complications in comparison to Conventional thyroidectomy technique.

ELIGIBILITY:
Inclusion Criteria:

* The limited size of the gland: volume less than 50 mm by ultrasound assessment. No evidence of retro-sternal extension. Benign nature of the disease proved by FNAC.

Exclusion Criteria:

* the patients who have one or more of the following criteria:

  1. The size of the gland is more than 50 mm by ultrasound assessment.
  2. Patients with retro-sternal goitre.
  3. Patients with proved malignancy or suspicious for malignancy by Ultrasonography(US) or by Fine-Needle Aspiration Cytology (FNAC).
  4. Previous surgery or radiotherapy to the neck.
  5. Thyroiditis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Degree of satisification of cosmetic appearance of the thyroidectomy scar | 12 months
  Degree of scar appearance satisification assessed by the patient and doctor using patient and observer scar assessment scale (POSAS) scale in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt